CLINICAL TRIAL: NCT02304224
Title: the Relationship of the Use of Eye Masks and Outcomes of Patients With Sepsis in Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Chen Yuanzhuo, M.D., Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 040114002
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Sepsis; Sleep Deprivation; Immune Suppression
Keywords: sepsis; melatonin; Human Leukocyte Antigen-DR; outcome
MeSH Terms: conditions — Sepsis; Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): the patients with sepsis admitted in the intensive care unit aren't applied with eye masks at night
- Eye masks (Experimental): the patients with sepsis in the intensive care unit are applied with eye masks at night in the duration of admission
  Interventions: Other: eye masks

INTERVENTIONS:
Other: eye masks — eye masks from 21:00 to 6:00 each night during admission
  Arms: Eye masks

SUMMARY:
The aim of the study is to investigate the relationship of nocturnal use of eye masks and immune function, cerebral function and outcomes of patients with sepsis. Thus more efficient and comprehensive treatment could be provided for patients in the duration of admission in intensive care unit.

DETAILED DESCRIPTION:
1. Treatment for patients There are no significant difference in standardized treatment received by patients enrolled, as well as the light equipment bedside and the food supply time. Patients are randomly divided into Eye Masks Group and Control Group by computer tools. Patients in Eye Masks Group are applied with eye masks from 22: 00 to 6: 00 each night during the admission. Blood sample was collected from each patient immediately after enrollment (D0), 6:30 of Day 1 (D1), Day 1 (D2), Day 3 (D3), Day 4 (D4) after admission. Urine of 6:00-21:00 and 21:00-6:00 is also stored from D0 to D4.
2. Clinical data collection Data such as patient's age, gender, contact information, time from onset to admission, existence of septic shock, pathogen species, the site of infection, the existence of organ dysfunction, APACHE II score (Acute Physiology And Chronic Health Evaluation Scoring System) , SOFA （Sequential Organ Failure Assessment）score, the use of mechanical ventilation, vasoactive drugs, corticosteroids, sedative and analgesic medication, history of eye diseases and neurological diseases is collected from each patient who is included in the study. Follow-up data for daily daytime sleep time, existence of delirium, CPC score and GCS score on Day 7 and Day 28, length of stay and survival of 28 days after admission is also collected.
3. Sample collection and processing The blood samples collected in citrate anticoagulation tubes and the urine samples collected in specialized graduated cylinders are stored at room temperature. Staining and fixation were performed within 24 h after blood collection. The expression of Monocyte Human Leukocyte Antigen-DR is detected using flow cytometer. The concentration of 6-sulfatoxymelatonin in urine is detected by ELISA kit.
4. Cerebral Performance Category (CPC) CPC is a 5-category scale for measuring neurological status 2 weeks after cardiac arrest and CPC score 6 months after cardiac arrest. The 5 categories are: CPC 1, conscious and alert with good cerebral performance; CPC 2, conscious and alert with moderate cerebral performance; CPC 3, conscious with severe cerebral disability; CPC 4, comatose or in persistent vegetative state; and CPC 5, brain dead, circulation preserved.
5. Glasgow Coma Scale (GCS) The GCS was developed as a standardized method for healthcare practitioners to evaluate degree of altered consciousness in patients who had sustained head injuries. The GCS is comprised of three categories: eye opening, verbal response, and motor response. The score from each category is summed, to provide a total GCS score (range 3-15).

ELIGIBILITY:
Inclusion Criteria:

1. Transferred into ICU before 21:00 the same day;
2. Consistent with the diagnosis of sepsis;
3. Written informed consent was obtained from patients or their family members.

Exclusion Criteria:

1. Age < 18 years;
2. With sleep disorders; mental illness; cancer; autoimmune diseases; dysfunction of liver or kidney;
3. History of using of immune-related drugs; melatonin receptor agonist or antagonist; sleep-aid or mental- related drugs;
4. History of accepting radiotherapy or chemotherapy;
5. Doing shift work before admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
survival of participants | up to 28 days after hospitalization

SECONDARY OUTCOMES:
Cerebral Performance Category（CPC) of Participants | up to 7 days after hospitalization
Cerebral Performance Category（CPC) of Participants | up to 28 days after hospitalization
Glasgow Coma Scale (GCS) of Participants | up to 7 days after hospitalization
Glasgow Coma Scale (GCS) of Participants | up to 28 days after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Yuanzhuo Chen, M.D., Study Chair — Shanghai 10th People's Hospital; Wenjie Li, M.D., Principal Investigator — Shanghai 10th People's Hospital; Huiqi Wang, M.D., Principal Investigator — Shanghai 10th People's Hospital; Chengjin Gao, M.D., Study Director — Shanghai 10th People's Hospital; Hu Peng, M.D., Study Director — Shanghai 10th People's Hospital; Yugang Zhuang, M.D., Principal Investigator — Shanghai 10th People's Hospital; Xiangyu Zhang, M.D., Study Director — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth Hospital, Shanghai, China